CLINICAL TRIAL: NCT02384785
Title: Effectiveness of Different Types of Therapeutic Currents in Clinical Dimension and Penetration Depth Dimension in Lower Back
Brief Title: Effectiveness of of Therapeutic Currents in Clinical Dimension and Penetration Depth Dimension in Lower Back
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-12-9941-IGA-CTIL
Record Dates: First submitted 2015-02-24; First posted 2015-03-10 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2016-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation; Transcranial Direct Current Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spinal Cord Stimulation: Patients who underwent implantation of electrodes spine for treatment in chronic pain.
  'Transcutaneous Electric Nerve Stimulation' and "Transcranial Direct Current Stimulation" (one after another)
  Interventions: Device: Transcutaneous Electric Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Electric Nerve Stimulation — Electric currents: 'Transcutaneous Electric Nerve Stimulation' and Transcranial Direct Current Stimulation will be applied on the back of the patients in parallel to the implanted electrodes. Implanted electrode will measure voltages that generated near the spinal cord tissue.
  Other Names: Transcranial Direct Current Stimulation

SUMMARY:
Electrical stimulation therapy for pain reduction was performed already 2000 years ago. In recent years many studies had proved the effectiveness of electrical stimulation in pain management, tissue healing and muscle strengthening. Today there are devices with many types of currents. Each current comes with different statements for its effectiveness and its penetration depth yet there is no consensus on the most effective current in the dimension of penetration depth.

DETAILED DESCRIPTION:
The study shall be recruited patients who underwent implantation of electrodes in the spine (Spinal Cord Stimulation- SCS). The electrode will serve as a voltage reader deep in the tissue. The voltage is generated from electrodes applied on the skin and delivers therapeutic currents to the patients back. The study will be tested 4 different types of currents and number of electrode placement.

ELIGIBILITY:
Inclusion Criteria:

* Normal cognitive status.
* language comprehension (understanding and speaking)a way that allows voluntary cooperation in research and compliance with the testing.

Exclusion Criteria:

* Pregnant women.
* neurological pathologies (such as -head injury) or other systemic diseases that affect the sensation (such as diabetes).
* Each participant which at any stage in research expresses his wish to resign.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who undergo electrodes implantation in lumbar spine due to chronic pain. Thease patients arrives 7 days after implantation to the clinic for a procedure of removing the electrodes.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2013-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The amount of electric voltage | monitoring voltage takes a few minutes only. Reading Voltage immidiatly- one test only for each current
  The amount of electric voltage generated by different types of currents and different electrodes locations

CONTACTS AND LOCATIONS:
Overall Officials: Moty Mr Ratmansky, MD, Study Chair — Site Sub-Investigator
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No